CLINICAL TRIAL: NCT05526781
Title: Visual Outcomes and Patient Satisfaction With Implantation of the Clareon Monofocal IOL With the New Clareon Manual Monarch IV IOL Delivery System
Status: Completed | Type: Observational
Sponsor: Eye Consultants of Atlanta (Other)
Collaborators: Sengi (Industry)
Responsible Party: Sponsor
Other Study IDs: JC-22-001
Record Dates: First submitted 2022-08-30; First posted 2022-09-02 (Actual); Results first posted 2025-03-26 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2025-03

CONDITIONS: Cataract
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- Clareon® monofocal Intraocular lens (toric and non-toric models): Bilateral implantation of the Clareon monofocal Intraocular lens (toric and non-toric models) with the Monarch IV inserter
  Interventions: Device: Clareon monofocal Intraocular lens (toric and non-toric models)

INTERVENTIONS:
Device: Clareon monofocal Intraocular lens (toric and non-toric models) — Bilateral implantation of the Clareon monofocal Intraocular lens (toric and non-toric models) with the Monarch IV inserter

SUMMARY:
To evaluate visual outcomes, in-the-bag placement and patient satisfaction in patients implanted with either Clareon monofocal or Clareon monofocal toric IOLs with the Monarch IV inserter and targeted for emmetropia.

DETAILED DESCRIPTION:
This study is a single-arm clinical evaluation study of visual performance and patient satisfaction, after successful bilateral cataract surgery. Subjects will be assessed pre- operatively, operatively and at 1 month and 3 months post-operatively. Clinical evaluations will include measurement of bilateral visual acuity, manifest refraction, and IOLSAT questionnaire.

ELIGIBILITY:
Inclusion Criteria:

Subjects are eligible for the study if they meet the following criteria: Note: Ocular criteria must be met in both eyes.

* Adult cataract surgical patients over the age of 45 with visually significant bilateral cataracts (glare visual acuity 20/40 or worse with BCVA testing), with planned cataract extraction using phacoemulsification, clear corneal incision and Clareon monofocal or Clareon toric with Monarch IV.
* Able to provide written informed consent for participation in the study.
* All eyes will be in the range of availability for Clareon monofocal and Clareon toric with Monarch IV.
* Expected visual potential of 20/25 Snellen (0.10 logMAR) or better in each eye.

Exclusion Criteria:

If any of the following exclusion criteria are applicable to the subject or either eye, the subject should not be enrolled in the study.

* Visually significant co-morbidities (corneal, retina, optic nerve disease) that could affect their satisfaction with surgery.
* History of neovascular AMD, diabetic macular edema, unstable proliferative diabetic retinopathy, geographic atrophy, branch retinal artery or branch retinal vein occlusion, central retinal artery or central retinal vein occlusion, moderate to severe epiretinal membrane, severe dry eye.
* History of intraocular infection including HSV keratitis, VZV keratitis, endophthalmitis.
* History of previous ocular surgery, including corneal refractive surgery, eye trauma or retinal detachment surgery.
* History of rheumatoid arthritis, ocular cicatricial pemphigoid, or Steven's Johnson Syndrome.
* History of glaucoma.

The principal investigator reserves the right to declare a patient ineligible or non- evaluable based on medical evidence that indicates they are unsuitable for the trial.

Pregnancy has a known effect on the stability of refractions and visual acuity. As such, subjects who become pregnant during the study will not be discontinued but their data may be excluded from analyses of effectiveness.

Min Age: 45 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Eligible participants will be presenting for cataract surgery and who are interested in and appropriate candidates for intraocular lens implantation.
Sampling Method: Non-Probability Sample
Enrollment: 34 (Actual)
Dates: Start 2022-09-21 (Actual); Primary Completion 2024-03-12 (Actual); Study Completion 2024-03-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joesph Christenbury, MD, Principal Investigator — Eye Consultants of Atlanta
Locations (1):
- Eye Consultants of Atlanta, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Clareon® Monofocal Intraocular Lens (Toric and Non-toric Models)
Started | 34
Completed | 33
Not Completed | 1
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Arm/Group | Clareon® Monofocal Intraocular Lens (Toric and Non-toric Models)
Number analyzed (Participants) | 28
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.6 (6.8)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Sex: Female | 13
  Sex: Male | 13
  Sex: Not Disclosed | 2
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Monocular Uncorrected Distance Visual Acuity (6m)
Time Frame: 3 months postoperative
Measure: Mean (Standard Deviation); unit: logMAR
Units Other Than Participants: eyes
Arm/Group | Clareon® Monofocal Intraocular Lens (Toric and Non-toric Models)
Number analyzed (Participants) | 28
Number analyzed (eyes) | 56
logMAR | 0.06 (0.07)

2. Primary Outcome: Binocular Uncorrected Distance Visual Acuity (6m)
Time Frame: 3 months postoperative
Measure: Mean (Standard Deviation); unit: logMAR
Arm/Group | Clareon® Monofocal Intraocular Lens (Toric and Non-toric Models)
Number analyzed (Participants) | 28
logMAR | 0.03 (0.04)

3. Primary Outcome: Binocular Corrected Distance Visual Acuity (6m)
Time Frame: 3 months postoperative
Measure: Mean (Standard Deviation); unit: logMAR
Arm/Group | Clareon® Monofocal Intraocular Lens (Toric and Non-toric Models)
Number analyzed (Participants) | 28
logMAR | 0.00 (0.02)

4. Primary Outcome: Monocular Corrected Distance Visual Acuity (6m)
Time Frame: 3 months postoperative
Measure: Mean (Standard Deviation); unit: logMAR
Units Other Than Participants: eyes
Arm/Group | Clareon® Monofocal Intraocular Lens (Toric and Non-toric Models)
Number analyzed (Participants) | 28
Number analyzed (eyes) | 56
logMAR | 0.00 (0.02)

5. Secondary Outcome: Monocular Uncorrected Intermediate Visual Acuity (66cm)
Time Frame: 3 months postoperative
Measure: Mean (Standard Deviation); unit: logMAR
Units Other Than Participants: eyes
Arm/Group | Clareon® Monofocal Intraocular Lens (Toric and Non-toric Models)
Number analyzed (Participants) | 28
Number analyzed (eyes) | 56
logMAR | 0.12 (0.05)

6. Secondary Outcome: Binocular Uncorrected Intermediate Visual Acuity (66cm)
Time Frame: 3 months postoperative
Measure: Mean (Standard Deviation); unit: logMAR
Arm/Group | Clareon® Monofocal Intraocular Lens (Toric and Non-toric Models)
Number analyzed (Participants) | 28
logMAR | 0.09 (0.05)

7. Secondary Outcome: Binocular Distance Corrected Intermediate Visual Acuity (66cm)
Time Frame: 3 months postoperative
Measure: Mean (Standard Deviation); unit: logMAR
Arm/Group | Clareon® Monofocal Intraocular Lens (Toric and Non-toric Models)
Number analyzed (Participants) | 28
logMAR | 0.0 (0.05)

8. Secondary Outcome: Monocular Distance Corrected Intermediate Visual Acuity (66cm)
Time Frame: 3 months postoperative
Measure: Mean (Standard Deviation); unit: logMAR
Units Other Than Participants: eyes
Arm/Group | Clareon® Monofocal Intraocular Lens (Toric and Non-toric Models)
Number analyzed (Participants) | 28
Number analyzed (eyes) | 56
logMAR | 0.05 (0.05)

9. Secondary Outcome: Manifest Refraction Spherical Equivalent (MRSE)
Description: The percentage of eyes with MRSE within ± 0.5 D.
Time Frame: 3 months postoperative
Measure: Count of Units; unit: eyes
Units Other Than Participants: eyes
Arm/Group | Clareon® Monofocal Intraocular Lens (Toric and Non-toric Models)
Number analyzed (Participants) | 28
Number analyzed (eyes) | 56
eyes | 51

10. Secondary Outcome: Overall Surgeon Satisfaction of Monarch IV Delivery Experience
Description: Score from 1-5. Higher scores indicate high surgeon satisfaction. Satisfaction was determined as the percentages of eyes where the surgeon was "Satisfied" or "Very Satisfied".
Time Frame: Operative visit (Day 0)
Measure: Count of Units; unit: eyes
Units Other Than Participants: eyes
Arm/Group | Clareon® Monofocal Intraocular Lens (Toric and Non-toric Models)
Number analyzed (Participants) | 28
Number analyzed (eyes) | 56
eyes | 56

11. Secondary Outcome: Consistency of In-the-bag Delivery of IOL During Implantation With Monarch IV
Description: Score from 1-4. Higher scores indicate higher consistency. Outcome measure is the percentage of eyes where the "IOL from cartridge coming out as planar, able to deliver IOL easily and smoothly into capsular bag".
Time Frame: Operative visit (Day 0)
Measure: Count of Units; unit: eyes
Units Other Than Participants: eyes
Arm/Group | Clareon® Monofocal Intraocular Lens (Toric and Non-toric Models)
Number analyzed (Participants) | 28
Number analyzed (eyes) | 56
eyes | 50

ADVERSE EVENTS:
Time Frame: 3 monts
Arm/Group | Clareon® Monofocal Intraocular Lens (Toric and Non-toric Models)
All-Cause Mortality (participants affected / at risk) | 0/28
Serious Adverse Events (participants affected / at risk) | 0/28
Other Adverse Events (participants affected / at risk) | 0/28

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-08-10): https://cdn.clinicaltrials.gov/large-docs/81/NCT05526781/Prot_SAP_000.pdf